CLINICAL TRIAL: NCT07210658
Title: Acceptability (Including Gastrointestinal Tolerance, Compliance and Palatability) of a Paediatric Oral Nutritional Supplement Containing Food Blends.
Brief Title: Acceptability, Gastrointestinal Tolerance, Compliance and Palatability Study.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ONS FB 001
Record Dates: First submitted 2025-07-23; First posted 2025-10-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Paediatrics
Keywords: Acceptability
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Children will act as their own control.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children will act as their own control for the nutritional product (Other)
  Interventions: Dietary Supplement: Oral nutritional supplementation

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplementation — As directed by the HCP

SUMMARY:
Acceptability, compliance and palatability study.

DETAILED DESCRIPTION:
Acceptability (including gastrointestinal tolerance, compliance and palatability) of a paediatric oral nutritional supplement containing food blends.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 1-15 years requiring 1 or more oral nutritional supplement to replace current oral nutritional supplement as part of their dietary management for disease related malnutrition.
* Patients well-established and stable on current nutritional support regimen.
* Willingly given, written, informed consent from patient/caregiver.

Exclusion Criteria:

* Unsafe swallow
* Inability to comply with the study protocol, in the opinion of the investigator.
* Under 1 years of age
* Patients on total parenteral nutrition
* Known food allergies, including any allergies to the ingredients
* Patients with Chronic Kidney Disease (CKD) stage 3b (G3b), stage 4 (G4), stage 5 (G5) or hepatic impairment.
* Participation in another interventional study within 2 weeks of this study.
* Patients with known or suspected ileus or mechanical bowel obstruction

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal tolerance | Days 1-7, and at day 14, 21 and 28
  Number of children who experienced gastrointestinal symptoms such as reflux, vomiting, nausea, constipation, diarrhoea recorded as a 4 point Likert scale as none, mild, moderate, severe symptoms at baseline and at post switch.

SECONDARY OUTCOMES:
Formula intake in mLs | 28 days
  The amount of mLs of formula intake by patient compared to what was prescribed in mLs.

CONTACTS AND LOCATIONS:
Locations (1):
- Dietetics, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided